CLINICAL TRIAL: NCT07395037
Title: Ward AdmiSsion of Haematuria: an Observational mUlticentre sTudy
Brief Title: A Study of Ward Admissions for Haematuria
Acronym: WASHOUT
Status: Recruiting | Type: Observational
Sponsor: British Urology Researchers in Surgical Training (Other)
Responsible Party: Sponsor
Other Study IDs: WASHOUT
Record Dates: First submitted 2025-03-14; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Urologic Diseases; Hematuria; Hematuria; Benign; Bladder Cancer; Renal Cancer; Urothelial Carcinoma
Keywords: catheter; haematuria; hematuria; irrigation
MeSH Terms: conditions — Urologic Diseases; Hematuria; Urinary Bladder Neoplasms; Kidney Neoplasms; Carcinoma, Transitional Cell | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective, obersational cohort (single cohort study): All patients meeting above defined inclusion and exclusion criteria. This study will take place in urological secondary and tertiary care centres internationally. The study will be conducted in centres that agree to participate in the study and meet the study's inclusion criteria below.
  Interventions: Other: Inpatient work-up and management

INTERVENTIONS:
Other: Inpatient work-up and management — The study hypothesis is that there is significant international and national variation in the diagnostic workup and management of patients requiring admission to the hospital with haematuria. Increased length of stay and poor outcomes in terms of mortality and healthcare costs are associated with management practices. The CRF will collect datapoints on inpatient work-up and management.

SUMMARY:
This multicenter, prospective observational study will evaluate national and international practice variations (if present) in the emergency management of patients admitted to hospital with haematuria, inform a consensus guideline for best practice and provide evidence to design an implementation study to optimise haematuria management pathway.

DETAILED DESCRIPTION:
The WASHOUT study is an international, multicentre prospective observational study designed to describe the management of patients with unplanned admission to hospital with haematuria. The study will utilise a collaborative methodology using the BURST model. Data on demographics, comorbidities, management practices, and outcomes will be collected using a standardised case report form and analysed using multilevel linear regression modelling. Primary outcomes include length of stay, while secondary outcomes cover diagnosis time, 90-day mortality, readmission rates, and resource use.

Patient and public involvement has been integral to the study design, ensuring that outcomes reflect patient priorities and that the research addresses key areas of concern

Study design and aim WASHOUT is an international, multicentre prospective observational study aiming to describe the management of haematuria emergency admissions.

Objectives:

Our objectives are:

Establish the incidence of causative diagnoses in patients being admitted with emergency haematuria.

Describe demographics, comorbidities, management and clinical outcomes of patients undergoing emergency admission to hospital with haematuria.

Identify factors associated with adverse outcomes and/or increased resource use.

Identify if variation in management and outcomes exists at local, regional and international levels.

Assess the impact different management pathways have on clinical outcomes (in terms of length of stay, health resource utilisation, readmission, 30-day and 90-day mortality rates Provide information to design a future randomised trial, for example control group outcomes and estimates of intra-cluster correlations.

Inclusion criteria Patients will be included consecutively if they are over 18 years of age and admitted to a participating secondary care centre as an emergency with haematuria under the primary or joint care of the urology team.

In the UK, individual consent is not necessary as this study has been considered a service evaluation.

Exclusion criteria any patients with catheter-related urethral trauma (defined as haematuria immediately after insertion of a urethral catheter without a preceding history of haematuria on this admission including traumatic catheter removal by patients), urological trauma (abdominal/pelvic) as well as patients who are in hospital less than 24 hours.

Primary outcome Length of stay, measured as the number of calendar days between the day of admission in the index hospital admission episode and the day of discharge from the hospital.

Secondary outcomes Time to definitive diagnosis measure, defined as the number of days between original presentation and final diagnosis.

30-day and 90-day mortality rate measured as the number of patients who died from the day of admission to the 30-day and 90-day follow-up period.

30-day and 90-day readmission rate, measured as the number of patients who were readmitted to the hospital with the same issue in the 30 days and 90-day after the date of discharge.

Number of days alive and out of hospital at 90 days. Healthcare costs, measured by calculating the cost of the stay, investigations, procedures, the patient underwent during the admission and in the 90-day follow-up period including readmissions.

The study will also assess current pathways that exist in hospitals, including acute care pathways and specific pathways for management of haematuria. Details will be obtained through a questionnaire distributed to each participating site.

Study delivery The study will utilise the The British Urology Researchers in Surgical Training (BURST) collaborative model. The design of the current study has been supported by input from the Centre for Healthcare Randomised Trials (CHaRT) (i.e. The Urology Foundation trials unit), who will be involved in designing and conducting the next study, which we anticipate will be an implementation randomised controlled trial.

Recruitment Patients will be recruited consecutively. The recruitment target for this study is based pragmatically on the prevalence of inpatient haematuria. Target recruitment per participating site is 15 patients across a 12-month period from 70 centres. The cumulative recruitment target from all sites is 1,050 patients. We want to recruit as many participants as possible during the 12-month period. The sample size is also based on the anticipated wide variation of practice and the heterogeneous nature of the presentation in terms of patient demographics and the underlying cause of the haematuria ranging from benign causes to malignant urological conditions. This sample size is also adequately powered to detect a meaningful difference in length of stay (defined as at least 1 day by study authors) using ANOVA to analyse any binary variable (spanning both clinicopathological features and management factors). This 1-day difference in length of stay is based on a calculated sample size of 1,054 patients, obtaining a power of 0.90 with a significance level of 0.05, and taking a standard deviation of length of stay as 5 days obtained from original data of a retrospective review covering this study population [2].

ELIGIBILITY:
Inclusion Criteria:

* Patients are included if they are over 16 years of age or older and admitted to a participating urological secondary care centre
* admitted as an emergency with haematuria as the primary or secondary diagnosis under the primary or joint care of urology

Exclusion Criteria:

* any patients under 16 years of age
* patients with catheter-related urethral trauma (defined as haemturia immediately after insertion of a urethral catheter that was documented as traumatic by the clinician, with no previous history of haemturia prior to catheter insertion)
* patients that are in hospital less than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included consecutively if they are over 18 years of age and admitted to a participating secondary care centre as an emergency with haematuria under the primary or joint care of the urology team.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Length of inpatient stay | At 90 days
  Number of calendar days between the day of admission in the index hospital admission episode and the day of discharge from the hospital.

SECONDARY OUTCOMES:
Mortality rate | At 90 days
Readmission rate | At 90 days
Time to definitive diagnosis | At 90 days
  Defined as the number of days between original presentation and final diagnosis.
Number of days alive and out of hospital | At 90 days.
  Composite endpoint - cumulative days alive and out of hospital
Resource use | At 90 days
  Calculating the cost of the inpatient stay, investigations, procedures, the patient underwent during the admission and in the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- BURST, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BURST website — https://www.bursturology.com/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT07395037/Prot_SAP_ICF_000.pdf